CLINICAL TRIAL: NCT06125912
Title: A Comparative Split-Face Study of the Effects of a Retinol Alternative Cream on Improving Facial Skin Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dime Beauty Co. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20361
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Arm (Experimental): All participants will use both the test product and the active control. Participants will use the creams in the evening, applying the TBT Cream to the right side of the face, and the positive control on the left side of the face.
  Interventions: Other: Dime Beauty TBT Cream; Other: Positive Control

INTERVENTIONS:
Other: Dime Beauty TBT Cream — Test product contains: Water, Ammonium Acryloyldimethyltaurate/VP Copolymer, Behenyl Alcohol, Dimethicone, Caprylic/Capric Tiglyceride, Cetearyl Alcohol, Dimethicone Crosspolymer, Glycerin, Glyceryl Stearate, Pentylene Glycol, 1,2-Hexanediol, Isododecane, Linoleic Acid, Caprylic/Capric/Succinic Triglyceride, Octadecene, Olea Europaea (Olive) Oil Unsaponifiables, Orobanche Rapum Extract, Phospholipids, Phytosterols, Polyglyceryl-6 Behenate, Polyglyceryl-6 Stearate, Propanediol, Pyrus Malus (Apple) Fruit Extract, Caprylic/Capric/Myristic/Stearic Triglyceride, Stearyl Dimethicone, Hydroxyacetophenone, Bakuchiol, Cetyl Ricinoleate, Tetrasodium Glutamate Diacetate, Tocopherol, Xanthan Gum.
Other: Positive Control — Water, Glycerin, Caprylic/Capric Triglyceride, Helianthus Annuus (Sunflower) Seed Oil, Pentylene Glycol, 1,2-Hexanediol, Cetearyl, Alcohol, Glyceryl Stearate, PEG-100 Stearate, Dimethicone, Hydroxyacetophenone, Sodium Ascorbate, Tocopherol, Carbomer, Xanthan Gum, Retinol, PEG-40 Hydrogenated Castor Oil.
  Other Names: 0.1% Retinol Clinical Trial Lotion

SUMMARY:
This study will evaluate the efficacy of the DIME TBT Cream in improving the appearance and hydration of aged skin in comparison to a retinol cream. This study will last for 60 days. The study will be conducted as a single-arm trial in which all participants will use both the test product and the positive control product (0.1% Retinol Clinical Trial Lotion). Participants will be required to undertake questionnaires at Baseline, Day 30, and Day 60. Photos will be taken at Baseline, Day 30, and Day 60, and expert skin grading will take place at Baseline and Day 60.

ELIGIBILITY:
Inclusion Criteria:

Females aged 18-65. Have one or more of the following: visible fine lines and wrinkles, dry skin, reduced skin elasticity, or generally unhealthy skin.

Must be willing to use two different skincare products, one on each side of their face for the duration of the trial.

Have a smartphone or camera to take before-and-after selfies.

Exclusion Criteria:

Anyone not in good health. Anyone who has any chronic health conditions such as oncological or psychiatric disorders.

Anyone who has any known serious allergic reactions that require the use of an Epi-Pen.

Anyone who is pregnant, breastfeeding, or wanting to become pregnant over the next three months.

Anyone who cannot/ will not commit to the study protocol. Anyone with a history of substance abuse.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Change in the appearance of fine lines and wrinkles on the face. [Baseline to Day 60] | 60 days
  Photos of the participants' face before and after the intervention will be evaluated for a change in this parameter by a board-certified dermatologist.
Change in participants' perception of the appearance of fine lines and wrinkles on the face. [Baseline to Day 60] | 60 days
  Measured via participant-reported questionnaires. Questionnaires will be designed using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Change in skin elasticity. [Baseline to Day 60] | 60 days
  Measured via participant-reported questionnaires. Questionnaires will be designed using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in signs of skin aging. [Baseline to Day 60] | 60 days
  Photos of the participants' face before and after the intervention will be evaluated for a change in this parameter by a board-certified dermatologist.
Changes in participants' perception of signs of skin aging. [Baseline to Day 60] | 60 days
  Measured via participant-reported questionnaires. Questionnaires will be designed using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in participants' perception of facial skin hydration. [Baseline to Day 60] | 60 days
  Measured via participant-reported questionnaires. Questionnaires will be designed using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in facial skin hydration. [Baseline to Day 60] | 60 days
  Photos of the participants' face before and after the intervention will be evaluated for a change in this parameter by a board-certified dermatologist.

SECONDARY OUTCOMES:
Comparison of the visual changes in the signs of skin aging as a result of using the test product compared to the control product. [Baseline to Day 60] | 60 days
  Photos of the participants' face before and after the intervention will be evaluated for a change in this parameter by a board-certified dermatologist. The left side of the face and the right side of the face will be compared.
Comparison of participants perception of the visual changes in the signs of skin aging as a result of using the test product compared to the control product. [Baseline to Day 60] | 60 days
  Measured via participant-reported questionnaires. Questionnaires will be designed using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe"). The left side of the face and the right side of the face will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided